CLINICAL TRIAL: NCT06508957
Title: Assessment of Sarcopenia and Bone Mineral Density Relation in Hip Fracture Patients: A Cross-Sectional Study by Using STAR Value
Brief Title: Sarcopenia and Bone Mineral Density Relation in Hip Fracture Patients
Status: Completed | Type: Observational
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Gamze Gul Gulec, DR, Kastamonu University
Other Study IDs: 2024-KAEK-26- 01
Record Dates: First submitted 2024-07-08; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Sarcopenia; Hip Fractures
Keywords: Sarcopenia; Hip Fractures; ultrasonic diagnosis
MeSH Terms: conditions — Sarcopenia; Hip Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hip fracture patients: this is a observational study. There is no intervention.

SUMMARY:
The study aims to investigate the relationship between sarcopenia and bone mineral density (BMD) in patients with hip fractures using sonographic thigh adjustment ratio (STAR) and dual-energy X-ray absorptiometry (DXA), as well as the relationship of sociodemographic factors, laboratory results, and comorbidities to these measurements.

Cross-sectional research was undertaken on patients with hip fractures in Kastamonu, Turkey. Sarcopenia was identified based on the ISarcoPRM algorithm, which utilizes poor grip strength (<22 kg for females and < 32 kg for males) along with low STAR values (< 1 for females and <1.4 for males). Sociodemographic data of the patients and levels of total protein, albumin, and 25-OH-vitamin D3 (25[OH]D) were obtained from all the patients. The BMD (bone mineral density) and T-scores of the proximal femur were measured using DXA (dual-energy X-ray absorptiometry).

DETAILED DESCRIPTION:
Introduction

Sarcopenia is a progressive and common skeletal muscle disorder, that causes progressive loss of age-related muscle strength and mass, associated with an increased likelihood of outcomes such as falls, fractures, physical disability, and death. Estimates place the overall prevalence of sarcopenia in older adults at approximately 10-40%. Osteoporosis and sarcopenia, prevalent conditions of advanced age, have comparable etiologies and risk factors. The co-occurrence of these illnesses amplifies the incidence of falls, fractures, and mortality. While EWGSOP2 and AWGS guidelines recommend using validated technologies like bioimpedance analysis, dual X-ray absorptiometry (DXA), computed tomography and magnetic resonance imaging for evaluating sarcopenia, these may not be feasible in certain clinical situations. The International Society of Physical and Rehabilitation Medicine (ISPRM) has suggested a different algorithm to diagnose sarcopenia by measuring anterior thigh muscle thickness using ultrasound (US). This method is easy to obtain, does not involve radiation, and is less expensive.

The study uses the sonographic thigh adjustment ratio (STAR) to look into the link between sarcopenia and bone mineral density (BMD) in people who have had a hip fracture. Additionally, the study explores the association between sociodemographic factors, laboratory results, comorbidities, and these measurements.

2. Material and Method

2.1. Study Design and Population

An observational cross-sectional study was conducted on hip fracture patients attending the orthopedic clinics of a tertiary hospital in Kastamonu, Turkey. The study was approved by the local Institutional Review Board (2024-KAEK-26- 01, February 7th, 2024). Written informed consent was obtained from all participants. Subjects were consecutively recruited during the first 24 hours of hospital stay from May to November 2023. Sarcopenia was diagnosed using the ISarcoPRM algorithm, which considers low grip strength and low STAR values. Inclusion criteria included the detection of low muscle strength with a hand dynamometer and patients scheduled for hip fracture surgery. Exclusion criteria included terminal disease, acute or chronic neuromuscular disease, and traumatic or pathological hip fracture.

2.2 Handgrip strength

Handgrip strength was measured using a Jamar dynamometer (Baseline Hydraulic Hand dynamometer, Irvington, NY) with participants performing two trials with both hands. The highest value obtained was used for analysis. Cut-off values for Turkish people were <22 kg for women and <32 kg for men.

2.3. Laboratory Data

The Kastamonu Research and Training Hospital Laboratory Service, a medical laboratory service with Turkey Accreditation System accreditation, performed laboratory analyses on-site. Total protein, albumin, and 25-OH-vitamin D3 (25[OH]D) levels were collected. The normal range for total protein is 6.6-8.3 g/dl, for albumin, it is 3.5-5.2 g/dl, and for 25[OH]D levels: deficient (<20 ng/dl), insufficient (20-30 ng/dl), or normal (>30 ng/dl).

2.4. Dual Energy X-ray Absorptiometry (DXA)

Non-fracture proximal femur neck BMD (g/cm2) and T-scores were obtained using the same DXA (Stratos DR (DMS) Mauguio, France). The World Health Organization (WHO) categorizes patients based on their lumbar spine, femoral neck, and/or total hip bone mineral density (BMD). Patients are classified as normal if their T score exceeds -1 standard deviation (SD), as osteopenic if it falls between -2.5 SD and -1 SD, and as osteoporotic if it equals or falls below - 2.5 SD. As only a small number of subjects presented with osteoporosis, "severe" osteopenia (-2.5 SD<T score ≤-2.0 SD) was added to the classification in our population.

2.5. Muscle Ultrasound(US) Measurements

Evaluation with the US (Mylab 25Gold, Esaote, Genova, Italy) was planned to be performed by the same clinicians using a 5-15 MHz linear probe in B mode, with the technique reported in previous studies. The thickness of the anterior thigh muscles was assessed in the non-fractured limb, between the anterior superior iliac spine and the proximal end of the patella with the patient lying in the supine position and the US probe placed perpendicularly with slight pressure. Once the muscle tissue was identified, the distance was measured between the femoral cortex and the most superficial muscle fascia (7). Measurements were obtained on two separate occasions by two different clinicians. The average value of a set of four consecutive measurements was calculated to assess the STAR value.

2.6. Sarcopenia Diagnosis

Sarcopenia was diagnosed according to the ISarcoPRM algorithm using low grip strength (< 22 kg for females and <32 kg for males) with low STAR values (<1 for females and <1.4 for males). The chair stand test, which is also recommended as a power and performance test to assess anterior thigh muscle function is unsuitable for this study's population with hip fractures. The STAR value was utilized to confirm the diagnosis. It is calculated by dividing the anterior thigh muscle thickness (mm) by the body mass value (kg/m2). According to prior research, the study used the established sonographic thigh adjustment ratio values of 1.0 for female patients and 1.4 for male subjects.

2.7. Statistical Analyses

Statistical analyses were performed with the SPSS v22 (SPSS Inc., Chicago, IL, USA) package. Quantitative data were summarized by mean ± standard deviation and median (minimum-maximum), while qualitative data were depicted as frequency and percentage. The Shapiro-Wilk test was performed to assess the normal distribution of the data, while the Levene test tested the homogeneity of variances. Two-sided independent t-tests were used to compare the mean for observations between sarcopenic and normal patients. Linear regressions and the Pearson coefficient were used to investigate associations and examine the relationship between parametric variables. Spearman's rho was used to investigate associations between nonparametric variables.

ELIGIBILITY:
Inclusion Criteria:

1. the detection of low muscle strength with a hand dynamometer
2. scheduled for hip fracture surgery.

Exclusion Criteria:

1. terminal disease
2. acute or chronic neuromuscular disease
3. traumatic or pathological hip fracture.

Ages: 58 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hip fracture patients attending the orthopedic clinics of a tertiary hospital in Kastamonu, Turkey.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density (g/cm2) | baseline
  Non-fracture proximal femur neck BMD (g/cm2) was obtained using the same DXA (Stratos DR (DMS), Mauguio, France)
Sonographic Thigh Adjustment Ratio (STAR) value | baseline
  The study used the standard sonographic thigh adjustment ratio values of 1.0 for female patients and 1.4 for male patients. These values are found by dividing the thickness of the anterior thigh muscle (in mm) by the person's body mass (in kg/m2).
T-scores | baseline
  A non-fracture proximal femur neck T score was obtained using the same DXA and is classified as normal if their T score exceeds -1 standard deviation (SD), as osteopenic if it falls between -2.5 SD and -1 SD, and as osteoporotic if it equals or falls below -2.5 SD.

SECONDARY OUTCOMES:
25[OH]D levels | baseline
Albumin levels | baseline
Protein levels | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Gamze Gül Güleç, Kastamonu, Turkey (Türkiye)

REFERENCES:
- [Background] Cruz-Jentoft AJ, Sayer AA. Sarcopenia. Lancet. 2019 Jun 29;393(10191):2636-2646. doi: 10.1016/S0140-6736(19)31138-9. Epub 2019 Jun 3. PMID 31171417
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Mayhew AJ, Amog K, Phillips S, Parise G, McNicholas PD, de Souza RJ, Thabane L, Raina P. The prevalence of sarcopenia in community-dwelling older adults, an exploration of differences between studies and within definitions: a systematic review and meta-analyses. Age Ageing. 2019 Jan 1;48(1):48-56. doi: 10.1093/ageing/afy106. PMID 30052707
- [Background] Teng Z, Zhu Y, Teng Y, Long Q, Hao Q, Yu X, Yang L, Lv Y, Liu J, Zeng Y, Lu S. The analysis of osteosarcopenia as a risk factor for fractures, mortality, and falls. Osteoporos Int. 2021 Nov;32(11):2173-2183. doi: 10.1007/s00198-021-05963-x. Epub 2021 Apr 20. PMID 33877382
- [Background] Gupta M, Lehl SS, Lamba AS. Ultrasonography for Assessment of Sarcopenia: A Primer. J Midlife Health. 2022 Oct-Dec;13(4):269-277. doi: 10.4103/jmh.jmh_234_22. Epub 2023 Apr 28. PMID 37324795
- [Background] Kara M, Kaymak B, Ata AM, Ozkal O, Kara O, Baki A, Sengul Aycicek G, Topuz S, Karahan S, Soylu AR, Cakir B, Halil M, Ozcakar L. STAR-Sonographic Thigh Adjustment Ratio: A Golden Formula for the Diagnosis of Sarcopenia. Am J Phys Med Rehabil. 2020 Oct;99(10):902-908. doi: 10.1097/PHM.0000000000001439. PMID 32941253
- [Background] Kara M, Kaymak B, Frontera W, Ata AM, Ricci V, Ekiz T, Chang KV, Han DS, Michail X, Quittan M, Lim JY, Bean JF, Franchignoni F, Ozcakar L. Diagnosing sarcopenia: Functional perspectives and a new algorithm from the ISarcoPRM. J Rehabil Med. 2021 Jun 21;53(6):jrm00209. doi: 10.2340/16501977-2851. PMID 34121127
- [Background] Bahat G, Tufan A, Tufan F, Kilic C, Akpinar TS, Kose M, Erten N, Karan MA, Cruz-Jentoft AJ. Cut-off points to identify sarcopenia according to European Working Group on Sarcopenia in Older People (EWGSOP) definition. Clin Nutr. 2016 Dec;35(6):1557-1563. doi: 10.1016/j.clnu.2016.02.002. Epub 2016 Feb 11. PMID 26922142
- [Background] Miron Mombiela R, Vucetic J, Rossi F, Tagliafico AS. Ultrasound Biomarkers for Sarcopenia: What Can We Tell So Far? Semin Musculoskelet Radiol. 2020 Apr;24(2):181-193. doi: 10.1055/s-0039-3402745. Epub 2020 May 21. PMID 32438444